CLINICAL TRIAL: NCT06834074
Title: Expanded Access Treatment of Neladalkib (NVL-655) in Patients With Advanced ALK+ NSCLC or Other ALK+ Solid Tumors
Brief Title: Expanded Access Program of Neladalkib (NVL-655) for Patients With Advanced ALK+ NSCLC or Other ALK+ Solid Tumors
Acronym: NVL-655-EAP
Status: Available | Type: Expanded Access
Sponsor: Nuvalent Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NVL-655-EAP
Record Dates: First submitted 2025-02-11; First posted 2025-02-19 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer; ALK-positive Non-small Cell Lung Cancer (NSCLC)
Keywords: ALK-positive Solid Tumors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: NVL-655 — Drug: NVL-655
  Other Names: Neladalkib

SUMMARY:
The Expanded Access Program will provide an alternate mechanism for patients, who lack satisfactory therapeutic alternatives and cannot participate in a neladalkib clinical trial, to access investigational neladalkib.

DETAILED DESCRIPTION:
The purpose of this Expanded Access Program is to provide investigational ALK inhibitor, neladalkib (NVL-655), for eligible patients with ALK-positive locally advanced or metastatic NSCLC (ALK+ NSCLC) who have previously received an ALK tyrosine kinase inhibitor (TKI) or eligible patients with other ALK-positive solid tumors, and lack satisfactory therapeutic alternatives and are unable to access neladalkib through a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Histologically or cytologically confirmed locally advanced or metastatic NSCLC or other solid tumors with a documented ALK rearrangement or activating ALK mutation.
3. Previously received at least one ALK TKI (for patients with NSCLC) or any prior therapy (for patients with other solid tumors), with no comparable or satisfactory alternative treatment options, in the opinion of the treating physician.
4. Enrollment in a clinical trial of neladalkib is not possible.
5. Adequate organ function and bone marrow reserve.

Exclusion Criteria:

1. Prior receipt of neladalkib.
2. Previous surgery, chemotherapy, radiotherapy or other anti-cancer therapy or participation in other studies within timeframe indicated in the protocol.
3. Ongoing anti-cancer therapy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (37):
- United States (11):
  - University Of California Irvine Medical Center, Orange, California
  - University of Colorado Anschutz School of Medicine, Aurora, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Cancer Institute, Detroit, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University, Durham, North Carolina
  - The Ohio State University, Columbus, Ohio
  - University of Washington / Fred Hutchinson Cancer Center, Seattle, Washington
- Australia (2):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer - Vancouver, Vancouver, British Columbia
  - Princess Margaret Hospital, Toronto, Ontario
- France (4):
  - Centre Leon Berard, Lyon, Auvergne-Rhône-Alpes
  - GCS IUCT Oncopole, Toulouse, Occitanie
  - CHU de Nantes, Nantes, Pays de la Loire Region
  - Institut Gustave Roussy, Villejuif, Île-de-France Region
- Netherlands (3):
  - Stichting Het Nederlands Kanker Instituut, Amsterdam, North Holland
  - Antoni van Leeuwenhoek Hospital, Amsterdam
  - University Medical Center Groningen, Groningen
- Singapore (2):
  - National University Hospital Singapore, Singapore
  - National Cancer Centre Singapore, Singapore
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea
- Spain (4):
  - Gerencia de Gestión Integrada A Coruna, A Coruña
  - Uomi Cancer Center-Clinica Tres Torres, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- Switzerland (2):
  - Kantonsspital Luzern, Lucerne
  - Ospedale Italiano di Lugano, Viganello
- Taiwan (2):
  - National Cheng-Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- United Kingdom (3):
  - The Royal Marsden Hospital, Sutton, Surrey
  - The Royal Marsden Hospital, London, UK
  - The Christie Hospital, Manchester